CLINICAL TRIAL: NCT00850096
Title: Effects of Nasulin v.Placebo on Blood Glucose Control in Patients With Type 2 DM Treated With Basal Insulin & Oral Antidiabetic Meds, Excluding Secretagogues in Phase 2A, Randomized, Parallel, Double-Blind, Placebo-Controlled, Multi-Center Study
Brief Title: Effects of Nasulin Versus Placebo on Blood Glucose Control in Patient Volunteers With Type 2 Diabetes Mellitus
Acronym: CPEX-011
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CPEX Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: US-0100-CPEX011
Record Dates: First submitted 2009-01-30; First posted 2009-02-24 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-11

CONDITIONS: Type 2 Diabetes
Keywords: Phase 2 Study for novel insulin delivery of type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo for Nasulin (Placebo Comparator): Placebo for Nasulin Spray
  Interventions: Other: Placebo for Nasulin
- Nasulin (Active Comparator): Nasulin (intranasal insulin spray 1%)
  Interventions: Drug: Nasulin

INTERVENTIONS:
Other: Placebo for Nasulin — Basal insulin (glargine) administered as a 1x daily injection in the morning and two placebo sprays administered three times daily just prior to meals for 6 weeks.
  Arms: Placebo for Nasulin
Drug: Nasulin — Basal insulin (glargine) administered as a 1x daily injection in the morning and two (50 IU) or four (100 IU) sprays of Nasulin (intranasal insulin spray 1%) administered three times daily just prior to meals for 6 weeks.
  Other Names: Intranasal insulin spray 1%
  Arms: Nasulin

SUMMARY:
The purpose of this study is:

* To assess the efficacy of Nasulin vs. placebo as indicated by time spent in euglycemia, assessed by continuous glucose monitoring data and serum fructosamine levels in patient volunteers with Type 2 Diabetes.
* To asses the safety and tolerability of Nauslin at 50 IU and 100IU doses in patient volunteers with Type 2 Diabetes

DETAILED DESCRIPTION:
This proof of concept trial has a randomized, parallel, double-blind, placebo-controlled design with a 4-week single-blind placebo and diet run-in period. Given a ratio of 1:1, patient volunteers will be randomized into one of two parallel treatment arms, Nasulin in a combination with insulin glargine or placebo in combination with insulin glargine. The randomization period will be 6 weeks in length. The total length of individual patient volunteer participation, including screening and follow-up will be approximately 13-14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Type 2 diabetes (18 years of age or older)
* Currently treated with basal insulin and OAD(s)
* HbA1c range of 6.5 - 10.
* BMI less than 41

Exclusion Criteria:

* Multiple daily injections of mealtime insulin
* Regular use of nasal sprays
* Significant nasal pathology
* Employed in a job which required irregular shift or night work

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Berman, MD, Study Director — CPEX Pharmaceuticals
Locations (21):
- United States (21):
  - Radiant Research, Chandler, Arizona
  - AMCR Institute, Inc, Escondido, California
  - Scripps Whittier Diabetes Clinic, La Jolla, California
  - Mills-Penninsula Health Services; Dorothy & Frank Diabetes Inst., San Mateo, California
  - Diablo Clinical Research, Walnut Creek, California
  - Barbara Davis Center, Aurora, Colorado
  - Clinical Research of West Florida, Clearwater, Florida
  - University of Miami Diabetes Research Institute, Miami, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - Maine Research Associates, Auburn, Maine
  - Washington University, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Mountain Diabetes and Endocrine Center, Asheville, North Carolina
  - ECU Diabetes Research Center, Greenville, North Carolina
  - Physician's East PA, Greenville, North Carolina
  - Texas Diabetes and Endocrinology, Austin, Texas
  - University of Texas; Southwestern Medical Center, Dallas, Texas
  - Rainier Clinical Research, Renton, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo for Nasulin | Nasulin
Started | 47 | 47
Completed | 44 | 45
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo for Nasulin | Nasulin | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (10.2) | 57.4 (8.85) | 56.3 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 18 | 45
  Male | 20 | 29 | 49
Region of Enrollment [Number; unit: participants]
  United States | 47 | 47 | 94

OUTCOME MEASURES:

1. Primary Outcome: Continuous Glucose Monitoring (CGM)
Description: Continuous glucose monitoring (CGM) data from patients receiving either Nasulin or placebo were collected and compared at baseline and the last two weeks of the study, and changes (week 5-6 minus baseline) in the mean percentage of time spend in euglycemia (70 to 180 mg/dl blood glucose) (MPTEU) were assessed from baseline Week 0 to Week 5-6.
Time Frame: Baseline and 5-6 weeks
Population: 47 patients were randomized to the placebo/oral antidiabetic arm while 47 others were randomized to the Nasulin/oral antidiabetic arm of the study. Forty-four patients in the placebo + oral antidiabetic arm and 45 patients in the Nasulin + oral antidiabetic arm completed the study.
Measure: Mean (Standard Error); unit: Percentage of day (24h) in euglycemia
Arm/Group | Placebo for Nasulin | Nasulin
Number analyzed (Participants) | 44 | 45
Percentage of day (24h) in euglycemia | -6.23 (3.295) | -0.72 (3.361)

2. Secondary Outcome: Overall Glycemic Control
Description: Continuous glucose monitoring (CGM) data from patients at the last weeks of study (week 5-6) were averaged for assessment of glycemic control under the treatment of either Nasulin or placebo.
Time Frame: 5-6 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Placebo for Nasulin | Nasulin
Number analyzed (Participants) | 44 | 45
mg/dl | 174.64 (3.962) | 163.34 (4.134)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Placebo for Nasulin | Nasulin
Serious Adverse Events (participants affected / at risk) | 3/47 | 2/47
Other Adverse Events (participants affected / at risk) | 35/47 | 28/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo for Nasulin (N=47) | Nasulin (N=47)
Abscess intra abdominal (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nasal irritation (General disorders) | 0 (0) | 1 (1)
Elevated blood cell count (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo for Nasulin (N=47) | Nasulin (N=47)
Ventricular tachychardia (Cardiac disorders) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0/0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 3 (3)
Ocular hyeraemia (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Application site irritation (General disorders) | 1 (1) | 4 (4)
Chest pain (General disorders) | 0 (0) | 1 (2)
Drug effect decreased (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 1 (1) | 3 (3)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 4 (4) | 0 (0)
Localized infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Confusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mucle strain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carotid bruit (Investigations) | 1 (1) | 0 (0)
Electrocadiogram abnormal (Investigations) | 1 (1) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremety (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (3)
Nasal congestion (Nervous system disorders) | 1 (1) | 2 (2)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Wheezing (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither the complete nor any part of the results of the study carried out under this protocol, nor any of the information provided by the sponsor for the purposes of performing the study, will be published or passed on to any third party without the consent of the study sponsor.